CLINICAL TRIAL: NCT06567821
Title: Using Navigation to Improve Accuracy of Maxillary Balloon Sinusotomy
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Dennis Tang, Physician, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: STUDY00003097
Record Dates: First submitted 2024-07-15; First posted 2024-08-23 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Chronic Maxillary Rhinosinusitis

STUDY DESIGN:
Intervention Model Description: This is a prospective randomized single blinded study. A block randomization will be performed to randomize each candidate to determine which side will receive a balloon sinusotomy without navigation and which side will receive balloon sinusotomy with the assistance of navigation. Each person has a set of sinuses on the right side and a set of sinuses on the left side. One side will be randomized to the balloon dilation with navigation while the other side will be performed with balloon dilation without navigation.
Who Masked: Outcomes Assessor
Masking Description: The procedure will be recorded for subsequent blinded review.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: RELIEVA SPINPLUS® NAV Balloon Sinusplasty System — The non-navigated device being used is the RELIEVA SPINPLUS® Balloon Sinusplasty System and the navigated device being used is the RELIEVA SPINPLUS® NAV Balloon Sinusplasty System. Both devices being used are standard devices that are currently FDA approved and used in practice for sinus dilation at Cedars-Sinai Medical Center.
  Other Names: RELIEVA SPINPLUS® Balloon Sinusplasty System

SUMMARY:
The purpose of the research is to examine the effectiveness of navigation in maxillary sinus balloon dilation for the treatment of chronic maxillary rhinosinusitis.

DETAILED DESCRIPTION:
The purpose of the research is to examine the effectiveness of navigation in maxillary sinus balloon dilation for the treatment of chronic maxillary rhinosinusitis. Adult patients (18 and over) with a confirmed diagnosis of chronic maxillary rhinosinusitis without nasal polyposis (CRSwNP) will undergo maxillary balloon sinusotomy. Block randomization will be performed to determine which side will receive balloon sinusotomy with navigation and which will have balloon sinusotomy using traditional anatomic landmarks. Participants will be followed for approximately 1 month post-procedure for a total study participation time of approximately 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older
* Candidate for primary endoscopic sinus surgery (ESS) for chronic maxillary rhinosinusitis without nasal polyposis (CRSwNP)
* Failed medical (non-surgical) therapy

Exclusion Criteria:

* History of previous sinus surgery
* Presence of nasal polyps
* Extensive sinonasal osteogeneis
* Cystic fibrosis
* Presence of sinonasal tumors
* Any records flagged "break the glass" or "research opt out."
* Any additional finding which in the opinion of the investigator precludes patient from participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Success Rate | 12 months
  There is a 30% expected improvement of success, in favor of navigation over non-navigation balloon sinuplasty devices.

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars Sinai, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided